CLINICAL TRIAL: NCT04149444
Title: A Phase 2 Study of Trifluridine/Tipiracil in Triple Negative Metastatic Breast Cancer
Brief Title: A Study of Trifluridine/Tipiracil in Triple Negative Metastatic Breast Cancer
Acronym: TACTIC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-103
Record Dates: First submitted 2019-10-23; First posted 2019-11-04 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARM 1 (Experimental): Dose escalation cohort - First 10 patients enrolled on study.
  Trifluridine/Tipiracil 30mg/m2 - to start, if no significant dose limiting side effects the dose will be increased to 35mg/m2 for the duration of the trial.
  After first 10 patients enrolled on study - Trifluridine/Tipiracil 35mg/m2
  Each cycle is 28 days. Two doses per day during days 1-5 with a two day rest for days 6 and 7. Then two doses per day for days 8-12, followed by a rest period for days 13-28 with the next cycle starting the day after day 28.
  Interventions: Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — Oral medication
  Other Names: TAS-102

SUMMARY:
This is an open-label, single arm, multi-stage, phase II trial of Trifluridine/tipiracil as a palliative treatment for patients with metastatic triple negative breast cancer who have failed both a taxane and anthracycline or have contraindications to these agents.

DETAILED DESCRIPTION:
This is an open-label, single arm, multi-stage, phase II trial of Trifluridine/tipiracil (TAS-102) as a palliative treatment for patients with metastatic triple negative breast cancer who have failed both a taxane and anthracycline or have contraindications to these agents.

The trial will begin with a safety run-in of 10 patients treated as follows:

Cycle 1: Trifluridine/tipiracil administered at 30 mg/m2 orally bid, 5 days per week, with 2 days of rest, for 2 weeks, followed by 14 day rest. Intra-patient dose escalation to 35 mg/m2 orally bid, 5 days per week, with 2 days of rest, for 2 weeks, followed by 14 day rest for subsequent cycles in the absence of dose limiting toxicities. As long as at least 80% of patients tolerate dose escalation, the trial will proceed to the next stage.

Patients enrolled in stages I and II will start Trifluridine/tipiracil at 35 mg/m2 orally bid, 5 days per week, with 2 days of rest, for 2 weeks, followed by 14 day rest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Life expectancy of ≥ 3 months
* Histologically or cytologically confirmed locally recurrent or metastatic breast cancer that is Estrogen receptor negative, Progesterone receptor negative, and HER2 normal on local testing
* Up to three prior chemotherapy regimens for advanced and/or metastatic disease
* Prior therapy with an anthracycline and a taxane in the adjuvant or metastatic setting or documented unsuitability
* Patients who developed advanced or metastatic disease within 6 months of completing adjuvant therapy are eligible with no prior therapy for advanced disease.
* Resolution of all chemotherapy- or radiation-related toxicities to ≤ grade 1 (except for stable sensory neuropathy ≤ grade 2 and alopecia) prior to commencement of study participation
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Adequate renal function: creatinine clearance ≥ 40 mL/min Cockcroft and Gault formula
* Adequate bone marrow function: absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, hemoglobin ≥ 10.0 g/dL (a hemoglobin <10.0 g/dL is acceptable if it is corrected by growth factor or transfusion), and platelet count ≥ 100 x 10^9/L
* Adequate liver function: bilirubin ≤ 1.5 times the upper limits of normal (ULN), alanine aminotransferase (ALT ≤ 3 x ULN (in the case of liver metastases ≤ 5 x ULN)
* Measurable disease (RECIST 1.1)
* Patients with known BRCA or ATM mutations or abnormalities (based on genomic profiling of tumor or germline genetic testing) are eligible if they meet all other inclusion criteria and have none of the exclusion criteria. The trial will not perform tumor genomic profiling or genetic testing but will document this information if available at study enrolment.
* Patients with known central nervous system (CNS) disease are eligible provided all of the following criteria are met:

  * Measurable disease outside the CNS
  * Metastases are limited solely to cerebellar and supratentorial lesions (i.e., no metastases to midbrain, pons, medulla, or spinal cord)
  * If corticosteroids are required, the patient must be on a stable dose or tapering dose of corticosteroids for 4 weeks prior to enrolment as therapy for CNS disease
  * Anticonvulsants at a stable dose are allowed as long as the patient has been seizure free for 3 weeks prior to enrolment
  * No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to randomization
  * No evidence of progression or haemorrhage after completion of CNS directed therapy
  * Note: Patients with new asymptomatic CNS metastases detected at the screening scan must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible, if all other criteria above are met.
* Women of child-bearing potential and males with female partners with child bearing potential must use highly effective contraceptive measures while taking Trifluridine/tipiracil and for 6 months after stopping treatment. Trifluridine/tipiracil may reduce the effectiveness of hormonal contraceptives, and therefore women using hormonal contraceptives should add a barrier contraceptive method.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to take and retain oral medications

Exclusion Criteria:

* Radiation therapy encompassing more than 30% of marrow
* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for at least 2 weeks prior to randomization.
* Leptomeningeal disease
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Trifluridine/tipiracil .
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because Trifluridine/tipiracil is an agent with the potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 8 weeks
  The Primary Endpoint ORR is calculated by taking the number of patients who at 8 weeks following initiation of Trifluridine/tipiracil have either a CR or a PR on first scan and dividing it over the total number of evaluable patients. Patients with stable disease are not included in this calculation.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 45 months.
  Progression free survival is defined as the time (in weeks) from the date of randomization until the date of the investigator-assessed radiological disease progression or death due to any cause. All patients will be followed until disease progression is documented according to RECIST 1.1 Criteria. The time measured in weeks between their baseline CT Scan and the first CT scan showing progressive disease as will be recorded as the progression free survival for that patient.
Disease Control Rate (DCR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 45 months.
  All patients who have either a Complete Response, Partial Response or exhibit stable disease for a minimum of 16 weeks will be counted as having achieved disease control. The number of patients attaining disease control will be divided by the total number of evaluable patients to attain a DCR for the entirety of the trial cohort.
Overall Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 45 months.
  The death of any patient in the trial from any cause will be recorded and the amount of time from enrollment in the trial until death will be recorded in weeks. A median overall survival for the entire cohort will then be calculated using this information.
Safety and Tolerability: All adverse events experienced by all patients | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 45 months.
  All adverse events experienced by all patients exposed to Trifluridine/tipiracil will be recorded and graded according to CTCAE version 5. These will be compared to the side effect profile presented in both the product monograph as well as the previously published phase III trial upon which the Health Canada approval is based.
Quality of Life - Using EQ5D - A standardized questionnaire measuring quality of life | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 32 months.
  Quality of life will be scored using the EQ5D. Patients will fill out this questionnaire prior to each follow up visit and the results will be compared within the same patient from visit to visit.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Tang, MD, Principal Investigator — Tom Baker Cancer Centre
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No